CLINICAL TRIAL: NCT05849194
Title: Role of Early Point of Care Ultrasound in Management of Sepsis in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0201798
Record Dates: First submitted 2023-04-26; First posted 2023-05-08 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2023-04

CONDITIONS: Sepsis
Keywords: Point of care ultrasound; Sepsis; Emergency department
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCUS group (Experimental): Group that will undergo POCUS examination
  Interventions: Diagnostic Test: POCUS examination
- Control group (No Intervention): The group that will not undergo POCUS examination

INTERVENTIONS:
Diagnostic Test: POCUS examination — Point of care ultrasound examination
  Arms: POCUS group

SUMMARY:
Aim of the study is to determine the diagnostic accuracy of point-of-care ultrasound and to determine its role in sepsis management .

DETAILED DESCRIPTION:
Two groups of patients will be studied one group will undergo POCUS examination and the other will not undergo POCUS examination then comparison between them will be done regarding accuracy of diagnosis and time taken to reach diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Emergency Department (ED) of Alexandria Main University Hospital (AMUH) with sepsis.
* Patients presented with septic shock.

Exclusion Criteria:

* Age less than 18
* Trauma patients.
* Pregnant females.
* Patients with terminal malignancy.
* Patients taking immunosuppressive drugs or chemotherapy.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of POCUS approach compared with the definitive diagnosis. | 8 months
  The study will include two groups of patients, POCUS group that will undergo point of care ultrasound (POCUS)examination in addition to clinical evaluation and laboratory investigations and control group that will not undergo POCUS examination but only undergo clinical evaluation and laboratory investigations. Both groups will be compared regarding proportion of accurate diagnosis (at emergency department)in relation to the final diagnosis that will be obtained after patient undergo further imaging techniques to search for sepsis such as chest X-ray or CT to look for chest infection and CT abdomen to confirm intra-abdominal sepsis.
  Unlike trauma, dyspnea and shock up till now there is no validated POCUS protocol to evaluate patients with sepsis.

SECONDARY OUTCOMES:
Time taken to reach diagnosis in both groups | 8 months
  Evaluation of the difference between two groups regarding time taken to reach diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria main university hospital, Alexandria, Egypt